CLINICAL TRIAL: NCT02008578
Title: Anti-Influenza Hyperimmune Intravenous Immunoglobulin Pilot Study (INSIGHT 005: Flu-IVIG Pilot)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14-I-0031; 14-I-0031
Record Dates: First submitted 2013-12-06; First posted 2013-12-11 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-08

CONDITIONS: Influenza
Keywords: Antiviral; Adjunctive Therapy; Antibody
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intravenous hyperimmune immunoglobulin (Flu-IVIG) (Experimental): Adults with confirmed Influenza A or B and evidence of ongoing viral replication (as demonstrated by positive rapid Ag or PCR preferably within 24 hours and no later than 6 days from symptom onset) will receive 0.25g Flu-IVIG/kg of actual body weight, to a maximum dose of 25g Flu-IVIG.
  Interventions: Biological: Intravenous hyperimmune immunoglobulin (Flu-IVIG)
- Placebo (Placebo Comparator): Adults with Influenza A or B and evidence of ongoing viral replication (as demonstrated by positive rapid Ag or PCR preferably within 24 hours and no later than 6 days from symptom onset) will receive placebo for Flu-IVIG (a comparable volume of saline).
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Intravenous hyperimmune immunoglobulin (Flu-IVIG)
  Arms: Intravenous hyperimmune immunoglobulin (Flu-IVIG)
Biological: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this randomized, double-blind, placebo-controlled trial of intravenous hyperimmune immunoglobulin (Flu-IVIG) in individuals with influenza A or B is to determine the pharmacokinetic (PK) profile of Flu-IVIG and assess whether antibody levels observed following Flu-IVIG transfusion are similar to those predicted. This pilot study will inform a larger study that will be powered to compare Flu-IVIG with placebo for efficacy.

DETAILED DESCRIPTION:
The purpose of this randomized, double-blind, placebo-controlled trial of intravenous hyperimmune immunoglobulin (Flu-IVIG) in individuals with influenza A or B is to determine the pharmacokinetic (PK) profile of Flu-IVIG and assess whether antibody levels observed following Flu-IVIG transfusion are similar to those predicted. This pilot study will inform a larger study that will be powered to compare Flu-IVIG with placebo for efficacy. In addition to informing the Flu-IVIG dosing required for the clinical outcomes trial, the pilot study will compare influenza antibody levels and safety for study participants randomly assigned Flu-IVIG and those assigned placebo, assess the feasibility of enrollment, evaluate randomization and blinding procedures, and possibly obtain some preliminary data on efficacy that may be used to inform sample size and study procedures for the clinical outcomes study.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Signed informed consent
  2. Age greater than or equal to 18 years of age
  3. Outpatients or inpatients who are PCR or rapid Ag positive for influenza A or B preferably within 24 hours and no later than 6 days from symptom onset
  4. Onset of illness no more than 6 days before randomization, defined as when the patient first experienced at least one respiratory symptom, constitutional symptom or fever
  5. For women of child-bearing potential, a negative pregnancy test within one day prior to randomization and a willingness to abstain from sexual intercourse or use at least 1 form of hormonal or barrier contraception through Day 28 of the study
  6. Willingness to have blood and respiratory samples obtained and stored

EXCLUSION CRITERIA:

1. If hospitalized, admitted for reasons other than influenza or complications of influenza
2. Women who are pregnant or breast-feeding
3. Strong clinical evidence (in the judgment of the site investigator) that the etiology of illness is primarily bacterial in origin.
4. Prior treatment with any investigational drug therapy within 30 days prior to screening
5. History of allergic reaction to blood or plasma products (as judged by the investigator)
6. Known IgA deficiency
7. A pre-existing condition or use of medication that, in the opinion of the investigator, may place the individual at a substantially increased risk of thrombosis (e.g., cryoglobulinemia, severe refractory hypertriglyceridemia, or clinically significant monoclonal gammopathy)
8. Serum creatinine greater than or equal to 1.5 x ULN or known active kidney disease that may affect drug pharmacokinetics (e.g., nephrotic syndrome)
9. Presence of any pre-existing illness that, in the opinion of the investigator, would place the individual at an unreasonably increased risk through participation in this study
10. Patients who, in the judgment of the investigator, will be unlikely to comply with the requirements of this protocol
11. Medical conditions for which receipt of 500mL volume may be dangerous to the patient (e.g., decompensated congestive heart failure)
12. Suspicion that infection is due to an influenza strain or subtype other than A(H1N1)pdm09, H3N2, or influenza B (e.g., H5N1, H7N9)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-12; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Hemagglutination Inhibition (HAI) titer for each influenza strain (H1N1, H3N2, B) taken 1 hour postinfusion compared to predicted levels. | 1 hour

SECONDARY OUTCOMES:
Compare HAI titers in active drug versus placebo recipients at 1 hour post-infusion, and Study Days 1, 3, and 7 according to the strain and subtype of virus with which participants are infected | Measured through Day 7
  assessment of influenza viral replication by Day 3; preliminary assessment of possible antiviral efficacy

OTHER OUTCOMES:
Length of hospital stay (for hospitalized participants) | Measured through the participant's hospital stay
Self-reported functional status and symptoms on Days 3 and 7 | Measured through Day 7
Adverse effects of the study treatment | Measured through Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Richard Davey, MD, Study Chair — National Institute of Allergy and Infectious Diseases (NIAID), NIH, Bethesda, MD 20892; Norman Markowitz, MD, Study Chair — The Henry Ford Hospital, Detroit, MI 48202
Locations (11):
- United States (11):
  - University of California at San Diego, San Diego, California
  - Denver Public Health, Denver, Colorado
  - George Washington University, Washington D.C., District of Columbia
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - Henry Ford Hospital, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Cooper University Hospital, Camden, New Jersey
  - Montefiore Medical Center, The Bronx, New York
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - University of Texas Southwestern Medical Center, Dallas, Texas

REFERENCES:
- [Background] Dwyer DE; INSIGHT Influenza Study Group. Surveillance of illness associated with pandemic (H1N1) 2009 virus infection among adults using a global clinical site network approach: the INSIGHT FLU 002 and FLU 003 studies. Vaccine. 2011 Jul 22;29 Suppl 2(0 2):B56-62. doi: 10.1016/j.vaccine.2011.04.105. PMID 21757105
- [Background] Luke TC, Kilbane EM, Jackson JL, Hoffman SL. Meta-analysis: convalescent blood products for Spanish influenza pneumonia: a future H5N1 treatment? Ann Intern Med. 2006 Oct 17;145(8):599-609. doi: 10.7326/0003-4819-145-8-200610170-00139. Epub 2006 Aug 29. PMID 16940336
- [Background] Perez-Padilla R, de la Rosa-Zamboni D, Ponce de Leon S, Hernandez M, Quinones-Falconi F, Bautista E, Ramirez-Venegas A, Rojas-Serrano J, Ormsby CE, Corrales A, Higuera A, Mondragon E, Cordova-Villalobos JA; INER Working Group on Influenza. Pneumonia and respiratory failure from swine-origin influenza A (H1N1) in Mexico. N Engl J Med. 2009 Aug 13;361(7):680-9. doi: 10.1056/NEJMoa0904252. Epub 2009 Jun 29. PMID 19564631
- [Derived] INSIGHT FLU005 IVIG Pilot Study Group. INSIGHT FLU005: An Anti-Influenza Virus Hyperimmune Intravenous Immunoglobulin Pilot Study. J Infect Dis. 2016 Feb 15;213(4):574-8. doi: 10.1093/infdis/jiv453. Epub 2015 Sep 15. PMID 26374911
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2014-I-0031.html